CLINICAL TRIAL: NCT00310180
Title: Program for the Assessment of Clinical Cancer Tests (PACCT-1): Trial Assigning Individualized Options for Treatment:The TAILORx Trial
Brief Title: Hormone Therapy With or Without Combination Chemotherapy in Treating Women Who Have Undergone Surgery for Node-Negative Breast Cancer (The TAILORx Trial)
Acronym: TAILORx
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: American College of Surgeons (Other); Cancer and Leukemia Group B (Network); NSABP Foundation Inc (Network); NCIC Clinical Trials Group (Network); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00707; NCI-2009-00707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-PACCT-1; 06-482; CDR0000472066; PACCT-1; PACCT-1 (Other: ECOG-ACRIN Cancer Research Group); PACCT-1 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH); NCT00554931 (obsolete NCT alias)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Breast Adenocarcinoma; Hormone Receptor Positive; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIB Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole; Radiotherapy; Radiation; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Oncotype DX recurrence score =< 10) (Experimental): Patients in this group receive hormone therapy with tamoxifen, anastrozole, letrozole, or exemestane PO for up to 5 years. Some patients then continue to receive hormone therapy for an additional 5 years.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Tamoxifen Citrate
- Group 2, Arm I (experimental) (Experimental): Patients receive hormonal therapy as in Group 1 at the discretion of the treating physician.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Drug: Tamoxifen Citrate
- Group 2, Arm II (standard) (Active Comparator): Patients receive standard combination chemotherapy at the discretion of the treating physician. Within 4 weeks after the last dose of chemotherapy, patients receive hormonal therapy as in Group 1 at the discretion of the treating physician.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Tamoxifen Citrate
- Group 3 (Oncotype DX recurrence score >= 26) (Experimental): Patients in this group receive combination chemotherapy followed by hormone therapy similar to the patients in group two who are assigned to receive both types of treatment.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; CGS-20267; CGS20267; Femara; Fempro
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy or partial breast irradiation
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group 1 (Oncotype DX recurrence score =< 10); Group 2, Arm II (standard); Group 3 (Oncotype DX recurrence score >= 26)
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI 46474; ICI-46474; ICI46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide

SUMMARY:
This randomized phase III trial studies the best individual therapy for women who have node-negative, estrogen-receptor positive breast cancer by using a special test (Oncotype DX), and whether hormone therapy alone or hormone therapy together with combination chemotherapy is better for women who have an Oncotype DX recurrence score of 11-25. Estrogen can cause the growth of breast cancer cells. Hormone therapy may fight breast cancer by blocking the use of estrogen by the tumor cells or by lowering the amount of estrogen the body makes. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving hormone therapy together with more than one chemotherapy drug (combination chemotherapy) has been shown to reduce the chance of breast cancer recurrence, but the benefit of adding chemotherapy to hormone therapy for women with node-negative, estrogen-receptor positive breast cancer is small. New tests may provide information about which patients are more likely to benefit from chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether adjuvant hormonal therapy is not inferior to adjuvant chemohormonal in women whose tumors meet established clinical guidelines for adjuvant chemotherapy and fall in the "primary study group" category (Oncotype DX Recurrence Score 11-25).

II. To create a tissue and specimen bank for patients enrolled in this trial, including formalin fixed paraffin embedded tumor specimens, tissue microarrays, plasma, and deoxyribonucleic acid (DNA) obtained from peripheral blood.

SECONDARY OBJECTIVES:

I. To determine whether adjuvant hormonal therapy is sufficient treatment (i.e. 10 year distant disease-free survival of at least 95%) for women whose tumors meet established clinical guidelines for adjuvant chemotherapy and who fall into the "Secondary Study Group-1" category (Oncotype DX Recurrence Score =< 10).

II. To compare the outcomes projected at 10 years by Adjuvant (with outcomes projected using classical pathologic information including tumor size, hormone receptor status, and histologic grade) with those made by the Genomic Health Oncotype DX test. Classical pathologic information and outcome results will also be used to create and refine models that would use classical information instead of or in combination with genomic tests.

III. To estimate failure rates as a function of recurrence score (RS) separately in the chemotherapy (arms C, D) and no chemotherapy (arms A, B) groups. The purpose of the analysis is to develop more precise estimates of the relationship between recurrence score and chemotherapy treatment effect, if any, at the upper range of the RS 11 - 25 group.

IV. To determine the prognostic significance of the Oncotype DX recurrence score and of the individual RS gene groups (proliferation gene group, human epidermal growth factor receptor [HER]2 gene group, estrogen receptor [ER] gene group, invasion gene group, and other genes).

TERTIARY OBJECTIVES:

I. To evaluate the effects of chemotherapy and hormonal therapy vs hormonal therapy alone on perceived cognitive impairment, fatigue, fear of recurrence among pre-menopausal patients, endocrine symptoms and sexual dysfunction, and overall health-related quality of life (HRQL).

II. To determine whether perceived cognitive impairment, fatigue, fear of recurrence, endocrine symptoms, and overall HRQL are similar for patients receiving chemotherapy plus hormonal therapy in secondary study group 2 as for those in the primary study group (arm D vs C).

III. To determine whether perceived cognitive impairment, fatigue, fear of recurrence, endocrine symptoms, and overall HRQL are similar for patients receiving hormonal therapy alone in secondary study group 1 as for those in the primary study group (arms A vs B).

IV. To determine whether age will be inversely associated with a fear of recurrence, independent of treatment assignment.

V. Among participants receiving hormonal treatment alone on arm A and arm B, to determine whether Oncotype DX Recurrence score will be inversely correlated with fear of recurrence.

VI. To create a biospecimen repository including plasma, serum and CellSearch cassettes containing circulating tumor cells (CTC) for evaluating determinants of late relapse, including candidate biomarkers reflecting occult tumor burden (e.g., CTCs and plasma tumor DNA) and host factors (e.g., estrogen, insulin growth factor-[IGF] axis, inflammation, etc).

VII. To create a biorepository of metastatic tumor samples in patients who have had a late relapse.

VIII. To determine body mass index (BMI) and comorbidity burden in patients with operable breast cancer five or more years after diagnosis.

IX. To determine whether there is a relationship between late relapse and BMI at diagnosis and at 5 years after diagnosis, and whether BMI-associated inflammatory and/or metabolic biomarkers are associated with early and late recurrence.

OUTLINE: This is a partially randomized study. Patients are assigned to 1 of 3 treatment groups.

GROUP 1 (SECONDARY STUDY GROUP 1; ONCOTYPE DX RECURRENCE SCORE [ODRS] =< 10): Patients receive standard hormonal therapy (e.g., tamoxifen alone orally (PO), aromatase inhibitor [e.g., anastrozole, letrozole, or exemestane] alone PO, or tamoxifen PO followed by aromatase inhibitor PO) at the discretion of the treating physician for 5 or 10 years.

GROUP 2 (PRIMARY STUDY GROUP; ODRS 11-25): Patients are randomized to receive either hormonal therapy alone or combination chemotherapy and hormonal therapy.

ARM I (EXPERIMENTAL): Patients receive hormonal therapy as in Group 1 at the discretion of the treating physician.

ARM II (STANDARD): Patients receive standard combination chemotherapy at the discretion of the treating physician. Within 4 weeks after the last dose of chemotherapy, patients receive hormonal therapy as in Group 1 at the discretion of the treating physician.

GROUP 3 (SECONDARY STUDY GROUP 2; ODRS >= 26): Patients receive combination chemotherapy as in Group 2, Arm II followed by hormonal therapy as in Group 1.

Patients in all groups who have had breast-conservation surgery are also treated with radiotherapy. Radiotherapy should begin within 4 weeks of registration for patients receiving hormonal therapy alone or within 8 weeks after completion of chemotherapy. Patients participating in National Surgical Adjuvant Breast and Bowel Project (NSABP) and/or Radiation Therapy Oncology Group (RTOG) partial irradiation trial(s) may receive partial breast radiation.

After completion of study treatment, patients are followed up every 3-6 months for 5 years and then annually for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable histologically confirmed adenocarcinoma of the female breast who have completed primary surgical treatment and meet the following criteria:

  * ER and/or progesterone receptor (PR)-positive: Estrogen and/or progesterone receptor positive disease (as defined by local pathology laboratory)
  * Negative axillary nodes: As assessed by a sentinel lymph node biopsy, an axillary dissection, or both, and as defined by the Sixth Edition of the American Joint Committee on Cancer (AJCC) staging criteria
  * Tumor size 1.1-5.0 cm (or 5 mm-1.0 cm plus unfavorable histological features):

    * Unfavorable features defined as intermediate or poor nuclear and/or histologic grade, or lymphovascular invasion
    * NOTE: Definition of tumor size: The tumor size used for determination of eligibility is the pathologic tumor size, which is usually determined by the size of the tumor as measured by inspection of the gross specimen; if the tumor size is measured microscopically and the tumor includes ductal carcinoma in-situ, the measurement should include only the invasive component of the tumor
  * The tumor must be human epidermal growth factor receptor 2 (Her2)/neu negative by either fluorescent in-situ hybridization (FISH) or immunohistochemistry (e.g. 0 or 1+ by DAKO Herceptest)
* The patient and physician must be agreeable to initiate standard chemotherapy and hormonal therapy as adjuvant therapy
* A tissue specimen from the primary breast cancer has been located and is ready to be shipped to the appropriate laboratory after consent is obtained and within 3 days following pre-registration; NOTE: For determination of the Oncotype Recurrence Score, tissue must be shipped to Genomic Health; if the Oncotype DX Recurrence Score was previously performed by Genomic Health (prior to pre-registration), tissue must be submitted to the Eastern Cooperative Oncology Group (ECOG)-American College of Radiology Imaging Network (ACRIN) Central Biorepository and Pathology Facility upon randomization
* Leukocyte count >= 3500/mm^3
* Platelets >= 100,000/mm^3
* Serum creatinine =< 1.5 mg/dL
* Serum aspartate transaminase (AST) that is =< 3-fold the upper institutional limits of normal
* Patients must be disease-free of prior invasive malignancies for >= 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix; patients with a previous ipsilateral or contralateral invasive breast cancer, or with bilateral synchronous cancers, are not eligible; patients with previous ipsilateral or contralateral ductal in situ carcinoma (DCIS) are not eligible
* Prior treatment

  * Mandatory prior surgery criteria:

    * Patient must pre-register within 84 days from the final surgical procedure required to adequately treat the primary tumor (please note that if margins are not clear and a resection has to be conducted after pre-registration but before randomization, the patient will be deemed to be within the 84 day window allowed by protocol and therefore eligible)
    * All tumors should be removed by either a mastectomy or local excision plus an acceptable axillary procedure (i.e., sentinel lymph node biopsy, axillary dissection, or both); there must be adequate (at least 1 mm if margin width specified) tumor-free margins of resection (for invasive and ductal carcinoma in-situ) in order for the patients to be eligible; patients with lobular carcinoma in-situ involving the resection margins are eligible
  * Criteria re: other prior treatments:

    * No prior chemotherapy for this malignancy
    * No prior radiation therapy for this malignancy; this includes no prior MammoSite Brachytherapy radiation therapy (RT)
    * Hormonal therapy: Patients who develop breast cancer while receiving a selective estrogen-receptor modulator (SERM; e.g., tamoxifen, toremifene, raloxifene) or an aromatase inhibitor (e.g., anastrazole, letrozole, exemestane) for breast cancer prevention or a SERM for other indications (e.g., raloxifene for osteoporosis) are not eligible; however, patients may have received up to 8 weeks of a SERM or aromatase inhibitor for this malignancy and still be eligible for study entry
* Patients must have an anticipated life expectancy of at least 10 years
* Patients with the following medical conditions should not be enrolled on the study:

  * Chronic obstructive pulmonary disease requiring treatment
  * Chronic liver disease (e.g., cirrhosis, chronic active hepatitis)
  * Previous history of a cerebrovascular accident
  * History of congestive heart failure or other cardiac disease that would represent a contraindication to the use of an anthracycline (e.g., doxorubicin or epirubicin)
  * Chronic psychiatric condition or other condition that would impair compliance with the treatment regimen
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to pre-registration to rule out pregnancy

  * Women of childbearing potential must be strongly advised to utilize an accepted and effective form of non-hormonal contraception (e.g. intrauterine device, condoms, diaphragm, abstinence)
* Patients must not have previously had the Oncotype DX Assay performed, with the exception of patients who have had the assay performed and have a recurrence score of 11-25

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10273 (Actual)
Dates: Start 2006-04-07 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2030-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Sparano, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1225):
- United States (1163):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Saint Bernards Regional Medical Center, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arroyo Grande Community, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - Community Cancer Institute, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - California Cancer Associates for Research and Excellence (cCare), Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Scripps Green Hospital, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Northridge Hospital Medical Center, Northridge, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Mercy Regional Cancer Center, Redding, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Breastlink Medical Group Inc, Santa Ana, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sansum Clinic Inc, Santa Barbara, California
  - Ray, Margaret, Savage. M.D. (UIA Investigator), Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Ridley-Tree Cancer Center-Solvang, Solvang, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Torrance Memorial Medical Center, Torrance, California
  - Emanuel Medical Center, Turlock, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - University of Connecticut, Farmington, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Harold Leever Regional Cancer Center, Waterbury, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Martin Medical Center, Stuart, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Martin Hospital South, Stuart, Florida
  - Space Coast Cancer Centers-Titusville, Titusville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - LaGrange Oncology Associates, Geneva, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Bloomington, Bloomington, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Research LLC, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - Medical Associates Clinic PC, Dubuque, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Metairie Oncologists, Metairie, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Overton Brooks Veteran's Administration Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - Mercy Hospital, Portland, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - York Hospital, York Village, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Commonwealth Hematology Oncology PC-Concord, Concord, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Dana Farber Community Cancer Care-Dorchester, Dorchester, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana Farber Community Cancer Care-Haverhill, Haverhill, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - HealthAlliance Hospital - Leominster, Leominster, Massachusetts
  - Saints Memorial Medical Center, Lowell, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Dana Farber Community Cancer Care-Stoneham, Stoneham, Massachusetts
  - Morton Hospital and Medical Center, Taunton, Massachusetts
  - Dana Farber Community Cancer Care-Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Reliant Medical Group Inc, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Crittenton Hospital, Rochester, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center, Jefferson City, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson-Tahoe Specialty Medical Center, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - John F Kennedy Medical Center, Edison, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Shore Memorial Hospital, Somers Point, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - San Juan Regional Medical Center, San Juan, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Catskill Regional Medical Center, Harris, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Queens Hospital Center, Jamaica, New York
  - Benedictine Hospital, Kingston, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - The Dyson Center for Cancer Care, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Highland Hospital, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moorehead Memorial Hospital, Eden, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Community Hospital and Wellness Centers, Bryan, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Stark, Michael, Edward. M.D. (UIA Investigator), Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Sky Lakes Medical Center - Cancer Treatment Center, Klamath Falls, Oregon
  - Asante Health System, Medford, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Conemaugh Memorial Medical Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple Health - Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Jones Clinic, Germantown, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - The Jackson Clinic PA, Jackson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Tennessee Oncology Elliston Place Plaza, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Thomas Midtown Hospital, Nashville, Tennessee
  - Saint Mary's North Cancer Center, Powell, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Texas Oncology Seton Northwest, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - The Center for Cancer and Blood Disorders-Burleson, Burleson, Texas
  - Texas Oncology-Cedar Park, Cedar Park, Texas
  - The Center for Cancer and Blood Disorders-Cleburne, Cleburne, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Dallas Oncology Consultants PA, Duncanville, Texas
  - The Center for Integrative Cancer Medicine, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - The Center for Cancer and Blood Disorders-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - The Center for Cancer and Blood Disorders-Mineral Wells, Mineral Wells, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology- San Marcos, San Marcos, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - The Center for Cancer and Blood Disorders-Weatherford, Weatherford, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Mount Ascutney Hospital and Health Center, Windsor, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Sentara Port Warwick, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Cancer Institutes of Washington PLLC, Yakima, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Surgical Associates Limited, Appleton, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Australia (14):
  - Border Medical Oncology, Albury, New South Wales
  - Coffs Harbour Health Campus-North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Lingard Private Hospital, Merewether, New South Wales
  - Royal Newcastle Hospital, Newcastle, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Nambour Hospital, Nambour, Queensland
  - Royal Hobart Hospital, Saint Hobart, Tasmania
  - Breast Unit-Mercy Private, East Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Saint John of God Hospital - Bunbury, Bunbury, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (27):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Health Sciences North, Greater Sudbury, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Trillium Health Partners - Queensway Health Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM-Hotel Dieu de Montreal, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Ireland (15):
  - Bon Secours Hospital, Cork, Co Cork
  - South Infirmary Victoria Hospital, Cork, Co Cork
  - Tallaght University Hospital, Dublin, Co Dublin
  - Saint Vincent's University Hospital, Dublin, Co Dublin
  - Mater Misericordiae University Hospital, Dublin, Co Dublin
  - Mater Private Hospital, Dublin, Co Dublin
  - Beaumont Hospital, Dublin, Co Dublin
  - Saint Vincent's Private Hospital, Mount Merrion, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
  - Mid-Western Regional Hospital, Limerick, Co Limerick
  - Sligo University Hospital, Sligo, Co Sligo
  - University Hospital Waterford, Waterford, Co Waterford
  - Cork University Hospital, Cork
  - Saint James Hospital, Dublin
  - Letterkenny General Hospital, Letterkenny
- New Zealand (3):
  - Auckland City Hospital, Grafton, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico
- Belfast City Hospital, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Derived] Kantor O, King TA, Freedman RA, Mayer EL, Chavez-MacGregor M, Korde LA, Sparano JA, Mittendorf EA. Racial and Ethnic Disparities in Locoregional Recurrence Among Patients With Hormone Receptor-Positive, Node-Negative Breast Cancer: A Post Hoc Analysis of the TAILORx Randomized Clinical Trial. JAMA Surg. 2023 Jun 1;158(6):583-591. doi: 10.1001/jamasurg.2023.0297. PMID 37043210
- [Derived] Sadigh G, Gray RJ, Sparano JA, Yanez B, Garcia SF, Timsina LR, Obeng-Gyasi S, Gareen I, Sledge GW, Whelan TJ, Cella D, Wagner LI, Carlos RC. Assessment of Racial Disparity in Survival Outcomes for Early Hormone Receptor-Positive Breast Cancer After Adjusting for Insurance Status and Neighborhood Deprivation: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Oncol. 2022 Apr 1;8(4):579-586. doi: 10.1001/jamaoncol.2021.7656. PMID 35175284
- [Derived] Yanez B, Gray RJ, Sparano JA, Carlos RC, Sadigh G, Garcia SF, Gareen IF, Whelan TJ, Sledge GW, Cella D, Wagner LI. Association of Modifiable Risk Factors With Early Discontinuation of Adjuvant Endocrine Therapy: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Oncol. 2021 Jun 17;7(8):1-7. doi: 10.1001/jamaoncol.2021.1693. Online ahead of print. PMID 34137783
- [Derived] Lynch SM, Russell NM, Barron S, Wang CA, Loughman T, Dynoodt P, Fender B, Lopez-Ruiz C, O'Grady A, Sheehan KM, Fay J, Amberger-Murphy V, Saha A, Klinger R, Gonzalez CA, Al-Attar N, Rahman A, O'Leary D, Lanigan FT, Bracken AP, Crown J, Kelly CM, O'Connor DP, Gallagher WM. Prognostic value of the 6-gene OncoMasTR test in hormone receptor-positive HER2-negative early-stage breast cancer: Comparative analysis with standard clinicopathological factors. Eur J Cancer. 2021 Jul;152:78-89. doi: 10.1016/j.ejca.2021.04.016. Epub 2021 Jun 2. PMID 34090143
- [Derived] Freidlin B, Hu C, Korn EL. Are restricted mean survival time methods especially useful for noninferiority trials? Clin Trials. 2021 Apr;18(2):188-196. doi: 10.1177/1740774520976576. Epub 2021 Feb 24. PMID 33626896
- [Derived] Wagner LI, Gray RJ, Sparano JA, Whelan TJ, Garcia SF, Yanez B, Tevaarwerk AJ, Carlos RC, Albain KS, Olson JA Jr, Goetz MP, Pritchard KI, Hayes DF, Geyer CE, Dees EC, McCaskill-Stevens WJ, Minasian LM, Sledge GW Jr, Cella D. Patient-Reported Cognitive Impairment Among Women With Early Breast Cancer Randomly Assigned to Endocrine Therapy Alone Versus Chemoendocrine Therapy: Results From TAILORx. J Clin Oncol. 2020 Jun 10;38(17):1875-1886. doi: 10.1200/JCO.19.01866. Epub 2020 Apr 9. PMID 32271671
- [Derived] Sparano JA, Gray RJ, Makower DF, Albain KS, Saphner TJ, Badve SS, Wagner LI, Kaklamani VG, Keane MM, Gomez HL, Reddy PS, Goggins TF, Mayer IA, Toppmeyer DL, Brufsky AM, Goetz MP, Berenberg JL, Mahalcioiu C, Desbiens C, Hayes DF, Dees EC, Geyer CE Jr, Olson JA Jr, Wood WC, Lively T, Paik S, Ellis MJ, Abrams J, Sledge GW Jr. Clinical Outcomes in Early Breast Cancer With a High 21-Gene Recurrence Score of 26 to 100 Assigned to Adjuvant Chemotherapy Plus Endocrine Therapy: A Secondary Analysis of the TAILORx Randomized Clinical Trial. JAMA Oncol. 2020 Mar 1;6(3):367-374. doi: 10.1001/jamaoncol.2019.4794. PMID 31566680
- [Derived] Korn EL, Gray RJ, Freidlin B. Noninferiority trials with nonadherence to the assigned randomized treatment. Clin Trials. 2019 Dec;16(6):673-681. doi: 10.1177/1740774519868479. Epub 2019 Aug 14. PMID 31409130
- [Derived] Sparano JA, Gray RJ, Ravdin PM, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Goetz MP, Olson JA Jr, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Berenberg JL, Abrams J, Sledge GW Jr. Clinical and Genomic Risk to Guide the Use of Adjuvant Therapy for Breast Cancer. N Engl J Med. 2019 Jun 20;380(25):2395-2405. doi: 10.1056/NEJMoa1904819. Epub 2019 Jun 3. PMID 31157962
- [Derived] Sparano JA, Gray RJ, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Goetz MP, Olson JA Jr, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Ravdin PM, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Berenberg JL, Abrams J, Sledge GW Jr. Adjuvant Chemotherapy Guided by a 21-Gene Expression Assay in Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):111-121. doi: 10.1056/NEJMoa1804710. Epub 2018 Jun 3. PMID 29860917
- [Derived] Sparano JA, Gray RJ, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Perez EA, Olson JA Jr, Zujewski J, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Ravdin P, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Atkins JN, Berenberg JL, Sledge GW. Prospective Validation of a 21-Gene Expression Assay in Breast Cancer. N Engl J Med. 2015 Nov 19;373(21):2005-14. doi: 10.1056/NEJMoa1510764. Epub 2015 Sep 27. PMID 26412349
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on April 7, 2006 and closed to registrations on October 6, 2010. A total of 11,232 patients were preregistered for Recurrence Score evaluation and 10,273 proceeded to register on the study.
Pre-assignment Details: Patients needed to be preregistered to the trial for ONCOTYPE recurrence score test, patients then were assigned or randomized to one of the four arms based on the recurrence score.
Groups:
- Arm A: Group 1 (Oncotype DX recurrence score =< 10): Patients in this group receive hormone therapy with tamoxifen, anastrozole, letrozole, or exemestane PO for up to 5 years. Some patients then continue to receive hormone therapy for an additional 5 years.
  Anastrozole: Given PO Exemestane: Given PO Letrozole: Given PO Tamoxifen: Given PO
- Arm B: Group 2 (Oncotype DX recurrence score 11-25): Patients receive hormone therapy with tamoxifen, anastrozole, letrozole, or exemestane PO for up to 5 years. Some patients then continue to receive hormone therapy for an additional 5 years.
  Anastrozole: Given PO Exemestane: Given PO Letrozole: Given PO Tamoxifen: Given PO
- Arm C: Group 2 (Oncotype DX recurrence score 11-25): Patients receive standard combination chemotherapy at the discretion of the treating physician. Within 4 weeks after the last dose of chemotherapy, patients receive hormonal therapy as in Group 1 at the discretion of the treating physician.
  Anastrozole: Given PO Exemestane: Given PO Letrozole: Given PO Tamoxifen: Given PO
  Combination chemotherapy: including oral CMF, IV CMF, standard AC, dose dense AC, standard AC-T, dose dense AC-T, FEC, TAC, TC, other protocol-specified regimens if participating in other CTSU trials including chemotherapy, and other regimens not protocol-specified if not participating in CTSU trials
- Arm D: Group 3 (Oncotype DX recurrence score >= 26): Patients in this group receive combination chemotherapy followed by hormone therapy similar to the patients in Group 2 who are assigned to receive both types of treatment.
  Anastrozole: Given PO Exemestane: Given PO Letrozole: Given PO Tamoxifen: Given PO
  Combination chemotherapy: including oral CMF, IV CMF, standard AC, dose dense AC, standard AC-T, dose dense AC-T, FEC, TAC, TC, other protocol-specified regimens if participating in other CTSU trials including chemotherapy, and other regimens not protocol-specified if not participating in CTSU trials
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 1629 | 3458 | 3449 | 1737
No On-study Data | 0 | 2 | 10 | 172
Ineligible | 3 | 4 | 6 | 7
No Follow-up Data | 7 | 55 | 131 | 245
Completed (Patients analyzed in the main analysis) | 1619 | 3399 | 3312 | 1389
Not Completed | 10 | 59 | 137 | 348

BASELINE CHARACTERISTICS:
Population: All eligible patients who had on-study data and follow-up data were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389 | 9719
Age, Customized [Count of Participants; unit: Participants]
  <=40 years | 58 | 154 | 157 | 79 | 448
  41-50 years | 371 | 985 | 920 | 330 | 2606
  51-60 years | 563 | 1235 | 1206 | 512 | 3516
  61-70 years | 518 | 868 | 895 | 395 | 2676
  71-75 years | 109 | 157 | 134 | 73 | 473
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1619 | 3399 | 3312 | 1389 | 9719
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 11 | 16 | 4 | 39
  Asian | 82 | 140 | 132 | 51 | 405
  Native Hawaiian or Other Pacific Islander | 8 | 7 | 14 | 1 | 30
  Black or African American | 107 | 236 | 235 | 115 | 693
  White | 1361 | 2883 | 2783 | 1162 | 8189
  More than one race | 2 | 5 | 2 | 1 | 10
  Unknown or Not Reported | 51 | 117 | 130 | 55 | 353
Recurrence score [Count of Participants; unit: Participants] — The Oncotype DX assay is a 21-gene assay that predicts the likelihood of chemotherapy benefit and 10-year risk of distant recurrence to inform adjuvant treatment decisions in certain women with early-stage invasive breast cancer. Oncotype DX test results assign a Recurrence Score, and the Oncotype DX Recurrence Score is a continuous score, ranged between 0 and 100, that provides an individual estimate of the 10 year risk of distant recurrence and predicts the likelihood of benefit from chemotherapy. Higher score indicate higher risk of recurrence.
  Participants
    0-5 | 432 | 0 | 0 | 0 | 432
    6-10 | 1187 | 0 | 0 | 0 | 1187
    11-15 | 0 | 1214 | 1159 | 0 | 2373
    16-20 | 0 | 1368 | 1344 | 0 | 2712
    21-25 | 0 | 817 | 809 | 0 | 1626
    26-30 | 0 | 0 | 0 | 598 | 598
    31-35 | 0 | 0 | 0 | 315 | 315
    36-40 | 0 | 0 | 0 | 158 | 158
    41-50 | 0 | 0 | 0 | 202 | 202
    >50 | 0 | 0 | 0 | 116 | 116

OUTCOME MEASURES:

1. Primary Outcome: 5-year Disease-free Survival
Description: Disease-free survival (DFS) is defined to be time from randomization to first event, where the first event is any of ipsilateral breast tumor recurrence, local recurrence, regional recurrence, distant recurrence, contralateral second primary invasive cancer, second primary non-breast invasive cancer (excluding non-melanoma skin cancers), or death without evidence of recurrence. The distribution of DFS (eg, 5-year DFS rate) is estimated using Kaplan-Meier method, and compared between the two randomized arms (arm B vs. arm C) using stratified log rank test and stratified Cox proportional hazard model.
Time Frame: Assessed every 6 months within 5 years from registration and then annually up to 20 years, DFS rate estimated at 5 years
Population: All eligible patients who had on-study data and follow-up data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389
percentage of participants | 94.0 [92.6 to 95.1] | 92.8 [91.8 to 93.6] | 93.1 [92.1 to 93.9] | 87.6 [85.5 to 89.4]
Statistical Analysis 1: Comparison: Arm B vs Arm C; This study uses a noninferiority design, but the noninferiority question is formulated using the conventional superiority null hypothesis of equal DFS on the two arms (that is, the null hypothesis is that Arm B is not inferior to Arm C). The alternative hypothesis is that Arm B has substantially worse DFS than Arm C, specified by a hazard ratio for B vs. C of 1.322; Test type: Superiority — Since the noninferiority comparison is formulated using a conventional superiority null hypothesis described as above, a type II error corresponds to concluding that Arm B is not inferior when in fact it is. The design therefore uses a one-sided type I error of 10% and is planned to have 95% power (5% type II error). If the null hypothesis is rejected (at the one-sided 10% level), then it will be concluded that endocrine therapy alone is inferior to chemoendocrine therapy; p = 0.13, Regression, Cox — One-sided p value for stratified Cox proportional hazard analysis, stratified on recurrence score, tumor size and menopausal status; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.94 to 1.24]

2. Secondary Outcome: 5-year Distant Recurrence-free Interval
Description: Distant recurrence-free interval (DRFI) is defined as time from date of randomization or registration to the date of distant recurrence of breast cancer, or of death with distant recurrence, if death is the first manifestation of distant recurrence. The distribution of DRFI (eg, 5-year DRFI rate) is estimated using Kaplan-Meier method.
Time Frame: Assessed every 6 months within 5 years from registration and then annually up to 20 years, DRFI rate estimated at 5 years
Population: All eligible patients who had on-study data and follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389
percentage of participants | 99.3 [98.8 to 99.6] | 98.0 [97.4 to 98.4] | 98.2 [97.6 to 98.6] | 93.0 [91.4 to 94.4]

3. Secondary Outcome: 5-year Recurrence-free Interval
Description: Recurrence-free interval (RFS) is defined as time from date of randomization or registration to the date of first recurrence of breast cancer (ipsilateral breast tumor recurrence, local/regional recurrence, distant recurrence) or to the date of death with recurrence, if death is the first manifestation of recurrence. The distribution of RFS (eg, 5-year RFS rate) is estimated using Kaplan-Meier method.
Time Frame: Assessed every 6 months within 5 years from registration and then annually up to 20 years, RFS rate estimated at 5 years
Population: All eligible patients who had on-study data and follow-up data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389
percentage of participants | 98.8 [98.1 to 99.2] | 96.9 [96.2 to 97.4] | 97.0 [96.3 to 97.6] | 91.0 [89.1 to 92.5]

4. Secondary Outcome: 5-year Overall Survival
Description: Overall survival (OS) is defined as time from date of randomization or registration to date of death from any cause. The distribution of OS (eg, 5-year OS rate) is estimated using Kaplan-Meier method.
Time Frame: Assessed every 6 months within 5 years from registration and then annually up to 20 years, OS rate estimated at 5 years
Population: All eligible patients who had on-study data and follow-up data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389
percentage of participants | 98.0 [97.2 to 98.6] | 98.0 [97.5 to 98.5] | 98.1 [97.6 to 98.5] | 95.9 [94.6 to 96.9]

5. Secondary Outcome: 5-year Disease-free Survival by Age and Recurrence Score Groups
Description: Disease-free survival (DFS) is defined to be time from randomization to first event, where the first event is any of ipsilateral breast tumor recurrence, local recurrence, regional recurrence, distant recurrence, contralateral second primary invasive cancer, second primary non-breast invasive cancer (excluding non-melanoma skin cancers), or death without evidence of recurrence. DFS is evaluated by recurrence score (0-10 vs. 11-15 vs. 16-20 vs. 21-25 vs. >25) and age groups (<=50 vs. 51-65 vs. 65-75). The distribution of DFS (eg, 5-year DFS rate) is estimated using Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All eligible patients who had on-study data and follow-up data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1619 | 3399 | 3312 | 1389
percentage of participants
  RS 0-10 & Age<=50 | 95.1 [92.4 to 96.8] | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A
  RS 0-10 & Age 51-65 | 94.7 [93.0 to 96.1] | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A
  RS 0-10 & Age 66-75 | 90.5 [86.5 to 93.3] | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A | NA [NA to NA] — Patients with RS of 0-10 were assigned to arm A
  RS 11-15 & Age <=50 | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C | 95.1 [92.5 to 96.8] | 94.3 [91.1 to 96.3] | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C
  RS 11-15 & Age 51-65 | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C | 95.5 [93.4 to 96.9] | 93.9 [91.7 to 95.6] | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C
  RS 11-15 & Age 66-75 | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C | 87.1 [80.9 to 91.4] | 91.4 [85.3 to 95.0] | NA [NA to NA] — Patients with RS of 11-15 were randomized to arm B or arm C
  RS 16-20 & Age <=50 | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C | 92.0 [89.0 to 94.2] | 94.7 [92.1 to 96.4] | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C
  RS 16-20 & Age 51-65 | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C | 94.3 [92.3 to 95.8] | 92.2 [89.9 to 94.0] | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C
  RS 16-20 & Age 66-75 | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C | 90.1 [84.6 to 93.8] | 90.2 [84.8 to 93.8] | NA [NA to NA] — Patients with RS of 16-20 were randomized to arm B or arm C
  RS 21-25 & Age <=50 | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C | 86.3 [81.1 to 90.2] | 92.1 [87.7 to 95.0] | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C
  RS 21-25 & Age 51-65 | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C | 91.6 [88.4 to 93.9] | 93.4 [90.5 to 95.4] | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C
  RS 21-25 & Age 66-75 | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C | 93.8 [87.9 to 96.8] | 90.9 [84.2 to 94.9] | NA [NA to NA] — Patients with RS of 21-25 were randomized to arm B or arm C
  RS >25 & Age <=50 | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | 86.4 [82.1 to 89.7]
  RS >25 & Age 51-65 | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | 87.5 [84.7 to 89.9]
  RS >25 & Age 66-75 | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | NA [NA to NA] — Patients with RS of >25 were assigned to arm D | 89.8 [84.4 to 93.4]
Statistical Analysis 1: Comparison: Arm B vs Arm C; Treatment interaction test was performed for the 9 age by RS subsets (3 groups for each, age groups <=50 vs. 51-65 vs. 66-75; RS groups 0-10 vs. 11-25 vs. >25) in patients randomized to arms B and C; Test type: Other — Treatment-by-Age and RS subset was performed via Cox proportional hazard analysis; p = 0.004, Regression, Cox

6. Secondary Outcome: To Compare the Outcomes Projected at 10 Years by Adjuvant! With Those Made by the Genomic Health Oncotype DX Test
Description: Adjuvant! is not currently available; additional work combining classical information with genomic tests will be reported separately.
Time Frame: Assessed at 10 years after study entry
Population: Outcome will never be analyzed.
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: 5-year Disease-free Survival by Individual RS Gene Groups
Description: Disease-free survival (DFS) is defined to be time from randomization to first event, where the first event is any of ipsilateral breast tumor recurrence, local recurrence, regional recurrence, distant recurrence, contralateral second primary invasive cancer, second primary non-breast invasive cancer (excluding non-melanoma skin cancers), or death without evidence of recurrence. The distribution of DFS (eg, 5-year DFS rate) is estimated using Kaplan-Meier method. 5-year DFS by individual RS gene groups (Proliferation Gene Group, HER2 Gene Group, ER Gene Group, Invasion Gene Group, and Other Genes) will be estimated in each arm.
Time Frame: Assessed every 6 months within 5 years from registration and then annually up to 20 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Both the chemotherapy and endocrine therapy given on this study were standard therapies for this population. To simplify the effort required for participating sites, adverse event data were not collected.
Description: Both the chemotherapy and endocrine therapy given on this study were standard therapies for this population. To simplify the effort required for participating sites, adverse event data were not collected.
Arm/Group | Arm A | Arm B | Arm C | Arm D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT00310180/Prot_SAP_000.pdf